CLINICAL TRIAL: NCT06634550
Title: Effect of Mulligan Technique Versus Core Stability Exercises on Low Back Pain in Post Menopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hala Ali Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005170
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mulligan technique group (Experimental): The participants will receive Mulligan technique and lifestyle modification advice for 4 weeks
  Interventions: Other: Mulligan technique; Other: Lifestyle modification advice
- Core stability exercise group (Experimental): The participants will receive core stability exercises and lifestyle modification advice for 4 weeks
  Interventions: Other: Core stability exercise; Other: Lifestyle modification advice
- Lifestyle modification advice group (Active Comparator): The participants will receive lifestyle modification advice only for 4 weeks
  Interventions: Other: Lifestyle modification advice

INTERVENTIONS:
Other: Mulligan technique — The participants will receive Mulligan technique (modified SNAGs) (10 rep. / 3 sets with 5 min rest in between) for 30 minutes, 3 sessions / week in addition to lifestyle modification advice for 4 weeks.
  Arms: Mulligan technique group
Other: Core stability exercise — The participants will perform core stability exercises (spinus multifiduse ex, diaphragmatic strengthening ex, frontal plank, pelvic floor ex,) 3 sessions / week for 30 min each session in addition to lifestyle modification advice for 4 weeks
  Arms: Core stability exercise group
Other: Lifestyle modification advice — The participants will receive lifestyle modification advice only for 4 weeks

SUMMARY:
This study will be conducted to compare the effect of Mulligan technique and core stability exercises on low back pain in post menopausal women.

DETAILED DESCRIPTION:
Low back pain is a major health problem affecting majority of the people at some point of their life.

Mulligan techniques can correct positional faults that occur in the spine and, thus, once the pain generator is released, normal function returns and the muscle guarding around the affected joint is resolved. Several studies have reported that along with the biomechanical changes, certain neurophysiological changes exist that occur at the spinal level after applying Mulligan techniques, including changes in descending pain inhibitory systems and changes in central pain processing mechanisms.

Core stability exercises are usually used to strengthen the muscles around the abdominal, lumbar, and pelvic regions, because the muscles of these regions play an important role in stability as well as in controlling the lumbar posture by using tonic or postural muscles during whole-body exercises.

So, this study will be conducted to provide new evidence and information about the efficacy of Mulligan technique versus core stability exercises on low back pain in postmenopausal women, to manage this problem for these women and add new information to the field of physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Sixty postmenopausal women (at least one year after stoppage of menses).
* Their age will be ranged from 50 to 60 years.
* All of them are diagnosed with chronic low back pain.
* Their BMI will be less than 30 kg/ m2.
* All of them are of sedentary lifestyle.
* The score of pain will be 2 or more in a VAS.

Exclusion Criteria:

* Participants will be excluded from the study if they have:
* Spinal fractures or any other neurological disorders.
* Lumber disc herniation or spondylolithesis
* Body mass index more than 30 kg/m2.
* Pelvic pathology
* Gynecological diseases as chronic pelvic pain, uterine prolapse or retroversion flexion of the uterus.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity level | 4 weeks
  The intensity of postmenopausal low back pain will be assessed using a visual analogue scale (VAS) for all participants in the three groups before and after treatment, which is a method of representing subjects' pain on a 10 cm linear scale. A score of 0 means " no pain" and 10 means " very high degree of pain
Lumbar flexion range of motion | 4 weeks
  The modified Schober test will be used to measure the lumbar flexion range of motion (ROM) by using the tape measurement. Each participant will be asked to stand erect with her feet about shoulder-width apart to stabilize the pelvis. Then, the posterior superior iliac spines(PSIS) will be determined by the therapist's both thumbs, and then an ink line will be drawn along the midline of the lumbar spines horizontal to the PSIS to mark the midpoint between the two PSIS. Then tape will be used to identify and mark two points: one is 10 cm superior to the midpoint (A), and another is 5 cm inferior to the midpoint (B). The participant will be instructed to bend forward as much as she can while keeping both knees straight, the new distance between superior and inferior skin marking will be measured in centimeters. The increased distance along the tape due to lumbar flexion is normally about 6-7 cm (less than 5 cm should be considered abnormal).
Lumbar extension range of motion | 4 weeks
  The modified Schober test will be used to measure the lumbar extension range of motion (ROM) by using the tape measurement while the patient is in a standing position. The participant will be instructed to put her hands on her buttocks and bend backward into full lumbar extension and the new distance between the superior and inferior skin markings will be measured in centimeters by the tape measurement. The change in the difference between the marks is used to indicate the amount of lumbar extension. The increased distance along the tape due to the extension of the lumbar spine is normally about 2-3 cm (less than 1cm should be considered abnormal).
Assessment of lateral flexion range of motion | 4 weeks
  The participant will be asked to stand erect with her feet about shoulder-width apart. Both right and left lateral flexion will be measured by the tape as the distance from the tip of the index finger to the floor at maximal comfortable lateral flexion. The participant will be instructed to bend her trunk laterally as much as she can. The normal value of lateral spinal flexion is 16.2-28.0 cm.

SECONDARY OUTCOMES:
Functional disability | 4 weeks
  Functional disability will be assessed by the Oswestry Disability Index, it was developed as clinical valid and reliable assessment tool that would provide an estimate of disability expressed as a percentage score. It is composed of 10 questions and it takes around 5min for a patient to complete. Each of the 10 questions is scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2. Scores are stratified into severity: 0-20, minimal disability; 21-40, moderate disability; 41-60, severe disability; 61-80, crippling back pain; 81-100, bed-bound. A low score = low degree of disability, a high score = high degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Azza B Kassab, professor, Study Chair — Cairo University
Locations (1):
- Hala Ali Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol